CLINICAL TRIAL: NCT02044055
Title: Hepatitis D Virus (HDV) Mother-To-Child Transmission (MTCT) From Hepatitis B Virus (HBV)-Hepatitis D Virus (HDV) Co-infected Pregnant Women: a Retrospective Study.
Brief Title: Mother-to-child Hepatitis D Transmission
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, Professor at University Paris VII Denis Diderot, physician, Hopital Lariboisière
Other Study IDs: Liver004
Record Dates: First submitted 2014-01-18; First posted 2014-01-23 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis D; Transmission
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children born to HBV-HDV women: Children born to HBV-HDV co-infected women will be checked for:
  * HDV antibodies
  * if positive, HDV RNA

SUMMARY:
HBV can be transmitted from mother-to-child, with a risk increasing according to maternal HBV DNA during pregnancy. HDV is a defective virus using HBs Ag for its own replication. Nucleosides analogues have only a minor impact on quantitative HBs Ag level. Data about vertical HDV transmission are old, justifying a new study.

DETAILED DESCRIPTION:
Hepatitis B Virus (HBV) can be transmitted from mother-to-child, with a risk increasing according to maternal HBV DNA viral load during the last trimester of pregnancy. Nucleosides analogues, lamivudine, telbivudine, or nucleotides analogues, tenofovir DF decrease HBV mother-to-child transmission risk, and are recommended in Guidelines (EASL 2012) for pregnant women with HBV DNA above 1,000 000 I.U/mL. HDV is a defective virus using HBs Ag for its own replication. HDV-HBV co-infection is a re-emerging infectious disease in western countries, due to immigration of people coming from endemic areas. Nucleosides analogues have only a minor impact on quantitative HBs Ag level (Boyd A et al. AIDS Research and Human Retroviruses 2013). Data about vertical HDV transmission are old (Rizzetto, et al. J Med Virol 1982), before a large use of nucleosides/nucleotides analogues in HBV infected pregnant women, justifying a new study.

ELIGIBILITY:
Inclusion Criteria:

* children born in the Maternity Department, Lariboisiere Hospital,
* from HBV-HDV co-infected women
* with a positive HDV RNA during pregnancy in the pregnant woman

Exclusion Criteria:

* negative HDV RNA during pregnancy in the pregnant woman

Ages: 9 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children born in the Maternity Department, Lariboisiere Hospital, from HBV-HDV co-infected women
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Hepatitis D antibodies (Ab) in children | up to 10 years (expected average: 5 years)
  Antibodies (Ab) against Hepatitis D Virus (HDV)

SECONDARY OUTCOMES:
HDV RNA in children with positive HDV Ab | up to 10 years (expected average: 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O SELLIER, M.D., Ph.D, Principal Investigator — Hopital Lariboisiere
Locations (1):
- Hopital Lariboisiere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sellier PO, Maylin S, Brichler S, Bercot B, Lopes A, Chopin D, Pogliaghi M, Munier AL, Delcey V, Simoneau G, Evans J, Gordien E, Simon F, Bergmann JF. Hepatitis B Virus-Hepatitis D Virus mother-to-child co-transmission: A retrospective study in a developed country. Liver Int. 2018 Apr;38(4):611-618. doi: 10.1111/liv.13556. Epub 2017 Sep 12. PMID 28834623